CLINICAL TRIAL: NCT05169931
Title: Clinical Efficacy of Amniotic Membrane Extract Eye Drops in Dry Eye Treatment
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding/support
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Saba K. Al-Hashimi, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-001915
Record Dates: First submitted 2021-12-14; First posted 2021-12-27 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Dry Eyes Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Treatment group to receive study drops (RegenerEyes) twice daily for 12 weeks
  Interventions: Biological: RegenerEyes

INTERVENTIONS:
Biological: RegenerEyes — Biologic eye drop

SUMMARY:
This prospective longitudinal study aims at evaluating the clinical efficacy of human amniotic fluid extract eye drops in the treatment of dry eye disease. 25 patients who are diagnosed with dry eye disease as defined by our criteria will be recruited from the cornea and dry eye clinic at Stein Eye Institute, UCLA. Pre-treatment baseline evaluations, 6 weeks, 12 weeks, and 24 weeks post treatment assessments will be performed by the principle investigator and co-investigator. All tests are considered non-invasive and are within the standard of practice in the evaluation for dry eye disease: (1) Ocular Surface Disease Index Questionnaire (OSDI); (2) Non-contact Tear Break-up Time (NITBUT); (3) Shirmer's test without anesthesia; (4) Ocular Surface Staining with Fluorescein and Lissamine green. Result of each test will be compared and analyzed to provide evidence of treatment efficacy. Treatment will be initiated for 12 weeks at a self-administered dose of one drop in both eyes two times per day. A follow-up of the study will be observed at the 24th week from the first day of treatment. All side effects and adverse events will be carefully observed and documented. Patients will be able to discontinue using the medication if they are not tolerating any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Presence of dry eye disease as defined as:

  1. Ocular Suface Disease Index (OSDI) score >13 AND EITHER i: Non-contact tear break-up time (NITBUT) < 10 seconds OR ii: Ocular Surface Staining (OSS) score > 1 in either eye

Exclusion Criteria:

1. Systemic diseases or comorbidities that may cause severe or secondary dry eye:

   1. Previous diagnosis of lymphoma, hepatitis C, HIV/AIDS, sarcoidosis, or amyloidosis that involves lacrimal glands
   2. Previous diagnosis of graft versus host disease (e.g., after bone marrow transplantation treatment for cancer) or cicatrizing conjunctivitis (e.g., Steven Johnson Syndrome, mucous membrane pemphigoid, trachoma)
   3. Anatomical or neurological lid closure problems (e.g., Bell's palsy, cicatricial ectropion, Alzheimer's disease, Parkinson's disease) 4
   4. Any history of chemotherapy, head or neck radiation treatment, or radioactive iodine treatment within 1 year prior to enrollment
   5. High dose oral or systemic steroids (equivalent to or greater than 5 mg prednisone) or immunosuppressive medication within 30 days prior to enrollment. Patients who are on stable dosing are eligible.
   6. Frequent or recent change in systemic medication regimen (e.g., diuretics, beta blockers, immunosuppressive medications, antidepressants that are known to interfere with dry eye) within 3 months prior to enrollment that may influence the ocular surface.
2. Other ocular surface diseases or surgical history that may cause severe or secondary dry eye:

   1. History of corneal dystrophy that in the opinion of the investigator is significantly affecting the ocular surface (e.g., significant anterior basement membrane dystrophy, Fuch's dystrophy with significant corneal edema and bullae, neurotrophic keratoconjunctivitis or corneal/conjunctival scarring including herpes simplex virus [HSV] or varicella zoster virus [VZV] keratitis)
   2. Any history of surgery for glaucoma (e.g., trabeculectomy, tube shunt)
   3. Corneal refractive surgery (e.g., laser in-situ keratomileusis [LASIK], photorefractive keratectomy [PRK], Intacs) within 6 months prior to enrollment
   4. Cataract, eyelid surgery, or retinal surgery (in operating room) within 6 months prior to enrollment
3. Use of treatments that may interfere with the ocular surface and/or treatment efficacy:

   1. Any in-office dry eye procedures (e.g., Intense Pulsed Light [IPL], LipiFlow®, nasolacrimal duct probing) within 30 days prior to enrollment
   2. Use of anti-glaucoma drops, topical antihistamines drops, or topical steroid drops within 7 days prior to enrollment
   3. Use of contact lenses. Patients willing to discontinue usage for 48 hours prior to each study visit will be eligible.
   4. Use of scleral lens, such as the prosthetic replacement of the ocular surface ecosystem (PROSE) lens
   5. Current use of topical lifitegrast (Xiidra®), topical cyclosporine (Restasis®), topical tacrolimus, or topical pimecrolimus. Patients willing to discontinue their due to insufficient benefit will be eligible.
4. Other important exclusion criteria:

   1. Current smoker (within 1 year prior to enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | 12 weeks
  Symptom Questionnaire

SECONDARY OUTCOMES:
Ocular Surface Staining Score | 12 weeks
Schirmer Score | 12 weeks
  Schirmer score after 5 minutes with anesthesia
Non-contact Tear Break-up Time | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Saba Al-Hashimi, M.D, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Neil EC, Henderson M, Massaro-Giordano M, Bunya VY. Advances in dry eye disease treatment. Curr Opin Ophthalmol. 2019 May;30(3):166-178. doi: 10.1097/ICU.0000000000000569. PMID 30883442
- [Background] Murri MS, Moshirfar M, Birdsong OC, Ronquillo YC, Ding Y, Hoopes PC. Amniotic membrane extract and eye drops: a review of literature and clinical application. Clin Ophthalmol. 2018 Jun 18;12:1105-1112. doi: 10.2147/OPTH.S165553. eCollection 2018. PMID 29950805
- [Background] Quinto GG, Camacho W, Castro-Combs J, Li L, Martins SA, Wittmann P, Campos M, Behrens A. Effects of topical human amniotic fluid and human serum in a mouse model of keratoconjunctivitis sicca. Cornea. 2012 Apr;31(4):424-30. doi: 10.1097/ICO.0b013e31823f0a64. PMID 22290385
- [Background] Yeu E, Goldberg DF, Mah FS, Beckman KA, Luchs JI, Solomon JD, White DE, Gupta PK. Safety and efficacy of amniotic cytokine extract in the treatment of dry eye disease. Clin Ophthalmol. 2019 May 27;13:887-894. doi: 10.2147/OPTH.S203510. eCollection 2019. PMID 31213759
- [Background] Chen M, Chang CK, Lin SY, Chen M. A Pilot Study of the Short Term Effectiveness and Safety of Amniotic Fluid in Severe Dry Eye Disease. Med Hypothesis Discov Innov Ophthalmol. 2019 Summer;8(2):81-84. PMID 31263717